CLINICAL TRIAL: NCT01423006
Title: Pilot Study on Focal Prostate Radio-Frequency Ablation for the Treatment of Very-Low Risk Prostate Cancer
Brief Title: Pilot Study on Focal Prostate Radio-Frequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Trod Medical, US,LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16584
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer
Keywords: Pilot; Ablation; Low Risk; Radio Frequency; RFA; minimally invasive; prostate gland
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Focal Prostate Radio-Frequency Ablation (Experimental): Treatment is performed under a spinal or general anesthetic and will include the one to three regions of the prostate containing cancer based on the mapping biopsy.
  Interventions: Procedure: Radio-Frequency Ablation (RFA) ENCAGE™

INTERVENTIONS:
Procedure: Radio-Frequency Ablation (RFA) ENCAGE™ — RFA is a minimally invasive procedure. It is an image-guided technique that heats and destroys cancer cells. In RFA, imaging techniques such as ultrasound or magnetic resonance imaging (MRI) are used to help guide a needle electrode into a cancerous tumor. High-frequency electrical currents are then passed through the electrode, destroying the cancer cells.
  Other Names: ENCAGE™

SUMMARY:
This is a prospective pilot study. The purpose of this research study is to evaluate the safety and efficacy of focal Radio-Frequency Ablation (RFA) in men with low-risk, clinically localized prostate cancer.

DETAILED DESCRIPTION:
RFA is a minimally invasive procedure. It is an image-guided technique that heats and destroys cancer cells. In RFA, imaging techniques such as ultrasound or magnetic resonance imaging (MRI) are used to help guide a needle electrode into a cancerous tumor. High-frequency electrical currents are then passed through the electrode, destroying the cancer cells. Use of an RFA device was approved by the Food and Drug Association (FDA) in 1997 for the purposes of treating soft tissue tumors. The device we (Moffitt Cancer Center) will be using in this study has clearance for clinical use from the FDA. The effectiveness of the device is measured using biopsy cores at the site of the cancer after the RFA procedure. To evaluate the benefits of this procedure, we will also evaluate the change in quality-of-life indicators from baseline to 6 months following RFA. RFA is being developed as a minimally invasive potential treatment for prostate cancer.

This research study is a pilot clinical trial. Pilot clinical trials are smaller versions of larger studies that are conducted to prepare for the larger study. This pilot study pre-tests a research device before a large-scale multicenter study is launched.

The specific purpose of this pilot trial is to find out if RFA can effectively treat prostate cancer with fewer side effects including effects on urination, bowel function, and sexual function. RFA for early stage prostate cancer is designed to affect only the part of the prostate where cancer has been detected. The reasoning for this approach is the smaller the area given RFA, the less damage to surrounding tissues.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate, confirmed by H.L. Moffitt Cancer Center review
* No prior treatment for prostate cancer including hormonal therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Prostate Cancer Clinical Stage T1c
* prostate-specific antigen (PSA) <10 ng/ml (this will be the PSA level prompting the initial prostate biopsy)
* Prostate size <60 cc on transrectal ultrasound
* If on anti-coagulation medications, must be able to suspend this therapy for a couple of weeks
* Adequate organ function Pre-enrollment biopsy parameters (as per H.L. Moffitt Cancer Center review)
* Minimum of 10 biopsy cores
* No biopsy Gleason grade 4 or 5
* Unilateral cancer (only right-sided or left-sided, not bilateral)
* No more than 50% cancer in any one biopsy core
* No more than 25% of cores containing cancer

Exclusion Criteria:

* Medically unfit for anesthesia
* Histology other than adenocarcinoma
* Biopsy does not meet inclusion criteria
* Men who have received any hormonal manipulation (antiandrogens; luteinizing hormone-releasing hormone (LHRH) agonist; 5-alpha-reductase inhibitors) within the previous 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Negative Prostate Biopsy Rate at Six Months | 6 Months
  The primary efficacy endpoint is negative biopsy rate at 6 months after focal bipolar RFA. Evaluable patients for this study will be those who complete up through the six month follow-up/evaluation procedure.

SECONDARY OUTCOMES:
Completion of Quality of Life (QOL) Assessment Questionnaires at Six Months | 6 Months
  Patients will complete the Expanded Prostate Cancer Index Composite (EPIC), American Urologic (AUA), Rectal Assessment Scale (RAS), and Sexual Health Inventory for Men (SHIM) questionnaires at baseline, 3 month and 6 month visits. QOL will be primarily based on the EPIC, developed to measure health related QOL among men with prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pow-Sang, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States